CLINICAL TRIAL: NCT06256614
Title: Washed Microbiota Transplantation for Type 1 Diabetes Mellitus: a Real World Research
Brief Title: Washed Microbiota Transplantation for Type 1 Diabetes Mellitus
Status: Recruiting | Type: Observational
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Other Study IDs: WMT-RWS-T1DM
Record Dates: First submitted 2024-01-27; First posted 2024-02-13 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Type 1 Diabetes
Keywords: washed microbiota transplantation; type 1 diabetes mellitus; glycemic variability; daily insulin dosage; hypoglycemia; insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fecal, urine, and blood samples before and after intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: WMT — Washed microbiota transplantation refers to the infusion of washed microbiota from healthy donor into patients' gastrointestinal tract. Participants will receive three doses of WMT for T1DM.

SUMMARY:
This is a real-world study to explore the safety and the efficacy of washed microbiota transplantation (WMT) for patients with Type 1 Diabetes Mellitus (T1DM).

DETAILED DESCRIPTION:
At least 20 subjects who meet all the inclusion criteria but do not meet any exclusion criteria will be enrolled in this study. Data of demographic characteristics, blood glucose fluctuation and variability, daily insulin dosage and clinical outcomes will be collected. After treatment, they will enter the follow-up period for safety and efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to enter the study:

1. At the time of informed consent, male or non-pregnant or non-lactating female.
2. The diagnostic criteria for T1DM are confirmed by previous medical record.
3. The subject or his/her legal representative gives informed consent, fully nderstands the purpose of the study, is able to communicate effectively with the investigator, and comprehends and complies with the requirements set forth in the study.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria must be excluded from the study:

1. Diagnosed as any type of diabetes other than type 1 diabetes mellitus;
2. Subjects with severe life-threatening complications diabetes (such as ketoacidosis, or acute coronary syndrome, etc.);
3. At the time of screening, the subject or his/her legal representative refuses to take effective contraception within 3 months after the last treatment.
4. According to the judgment of the investigator, the subjects are not suitable to participate in this clinical study, or participation in this clinical study cannot guarantee the rights and interests of the subjects.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: National patients with T1DM receiving WMT will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
The mean daily insulin dosage of participants | One-week, Two-week, Four-week post-WMT
  The mean daily insulin dosage of participants in past week

SECONDARY OUTCOMES:
The Blood glucose of Time in Range (TIR, percent) of type 1 diabetes mellitus. | One-week, Two-week, Four-week post-WMT
  The proportion of time spent within the target blood sugar range (typically 3.9 to 10.0mmol/L) over a 24-hour period
The SD of blood glucose (SDBG, mmol/L) of type 1 diabetes mellitus. | One-week, Two-week, Four-week post-WMT
  The standard deviation of measured values during immediate blood glucose monitoring
The largest amplitude of glycemic excursions (LAGE, mmol/L) of type 1 diabetes mellitus. | One-week, Two-week, Four-week post-WMT
  The range of blood glucose values observed during immediate blood glucose monitoring
The mean amplitude of glycemic excursion (MAGE, mmol/L) of type 1 diabetes mellitus. | One-week, Two-week, Four-week post-WMT
  After filtering out blood glucose fluctuations below a certain threshold (usually 1 SD), the average fluctuation amplitude is calculated based on the direction of the first significant fluctuation
The mean of daily differences (MODD, mmol/L) of type 1 diabetes mellitus. | One-week, Two-week, Four-week post-WMT
  The average absolute difference between corresponding measured values over a continuous 48-hour period
The postprandial glucose excursions (PPGE, mmol/L) of type 1 diabetes mellitus. | One-week, Two-week, Four-week post-WMT
  The average absolute difference between post-meal blood glucose taken 2 hours after three meals and the corresponding pre-meal blood glucose.
The mean blood glucose (MBG, mmol/L) of type 1 diabetes mellitus. | One-week, Two-week, Four-week post-WMT
  Average values obtained from immediate blood glucose monitoring
The coefficient of variation (CV, percent) of type 1 diabetes mellitus. | One-week, Two-week, Four-week post-WMT
  CV=(SDBG÷MBG)×100%
The frequency of hypoglycemia or duration of hypoglycemic state in the last 1 week | One-week, Two-week, Four-week post-WMT
  Hypoglycemia is defined as blood glucose < 3.9 mmol/L
The islet β-cell function after WMT compared with baseline | Three-day, One-week, Two-week, Four-week post-WMT
  2-hour postprandial C-peptide release was used to reflect islet β-cell function
The incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0 | One-week, Two-week, Four-week post-WMT
  The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang L, Peng W, Zhao Z, Zhang M, Shi Z, Song Z, Zhang X, Li C, Huang Z, Sun X, Wang L, Zhou M, Wu J, Wang Y. Prevalence and Treatment of Diabetes in China, 2013-2018. JAMA. 2021 Dec 28;326(24):2498-2506. doi: 10.1001/jama.2021.22208. PMID 34962526
- [Background] Li Y, Teng D, Shi X, Qin G, Qin Y, Quan H, Shi B, Sun H, Ba J, Chen B, Du J, He L, Lai X, Li Y, Chi H, Liao E, Liu C, Liu L, Tang X, Tong N, Wang G, Zhang JA, Wang Y, Xue Y, Yan L, Yang J, Yang L, Yao Y, Ye Z, Zhang Q, Zhang L, Zhu J, Zhu M, Ning G, Mu Y, Zhao J, Teng W, Shan Z. Prevalence of diabetes recorded in mainland China using 2018 diagnostic criteria from the American Diabetes Association: national cross sectional study. BMJ. 2020 Apr 28;369:m997. doi: 10.1136/bmj.m997. PMID 32345662
- [Background] Guideline for the prevention and treatment of type 2 diabetes mellitus in China (2020 edition)(Part 1). Chinese Journal of Practical Internal Medicine. 2020;41(8):668-695.
- [Background] Guideline for the prevention and treatment of type 2 diabetes mellitus in China (2020 edition)(Part 2). Chinese Journal of Practical Internal Medicine. 2020;41(9):757-784.
- [Background] Liu J, Liu M, Chai Z, Li C, Wang Y, Shen M, Zhuang G, Zhang L. Projected rapid growth in diabetes disease burden and economic burden in China: a spatio-temporal study from 2020 to 2030. Lancet Reg Health West Pac. 2023 Feb 3;33:100700. doi: 10.1016/j.lanwpc.2023.100700. eCollection 2023 Apr. PMID 36817869
- [Background] Zhong VW, Yu D, Zhao L, Yang Y, Li X, Li Y, Huang Y, Ding G, Wang H. Achievement of Guideline-Recommended Targets in Diabetes Care in China : A Nationwide Cross-Sectional Study. Ann Intern Med. 2023 Aug;176(8):1037-1046. doi: 10.7326/M23-0442. Epub 2023 Aug 1. PMID 37523704
- [Background] Experts consensus on management of glycemic variability of diabetes mellitus. Chin J Endocrinol Metab. 2017;33(8):633-636.
- [Background] Coutinho M, Gerstein HC, Wang Y, Yusuf S. The relationship between glucose and incident cardiovascular events. A metaregression analysis of published data from 20 studies of 95,783 individuals followed for 12.4 years. Diabetes Care. 1999 Feb;22(2):233-40. doi: 10.2337/diacare.22.2.233. PMID 10333939
- [Background] Su G, Mi S, Tao H, Li Z, Yang H, Zheng H, Zhou Y, Ma C. Association of glycemic variability and the presence and severity of coronary artery disease in patients with type 2 diabetes. Cardiovasc Diabetol. 2011 Feb 25;10:19. doi: 10.1186/1475-2840-10-19. PMID 21349201
- [Background] Su G, Mi SH, Tao H, Li Z, Yang HX, Zheng H, Zhou Y, Tian L. Impact of admission glycemic variability, glucose, and glycosylated hemoglobin on major adverse cardiac events after acute myocardial infarction. Diabetes Care. 2013 Apr;36(4):1026-32. doi: 10.2337/dc12-0925. Epub 2013 Jan 24. PMID 23349547
- [Background] Jin SM, Kim TH, Oh S, Baek J, Joung JY, Park SM, Cho YY, Sohn SY, Hur KY, Lee MS, Lee MK, Kim JH. Association between the extent of urinary albumin excretion and glycaemic variability indices measured by continuous glucose monitoring. Diabet Med. 2015 Feb;32(2):274-9. doi: 10.1111/dme.12607. Epub 2014 Oct 29. PMID 25307609
- [Background] Hsu CR, Chen YT, Sheu WH. Glycemic variability and diabetes retinopathy: a missing link. J Diabetes Complications. 2015 Mar;29(2):302-6. doi: 10.1016/j.jdiacomp.2014.11.013. Epub 2014 Dec 3. PMID 25534877
- [Background] Surawicz CM, Brandt LJ, Binion DG, Ananthakrishnan AN, Curry SR, Gilligan PH, McFarland LV, Mellow M, Zuckerbraun BS. Guidelines for diagnosis, treatment, and prevention of Clostridium difficile infections. Am J Gastroenterol. 2013 Apr;108(4):478-98; quiz 499. doi: 10.1038/ajg.2013.4. Epub 2013 Feb 26. PMID 23439232
- [Background] Sampson TR, Debelius JW, Thron T, Janssen S, Shastri GG, Ilhan ZE, Challis C, Schretter CE, Rocha S, Gradinaru V, Chesselet MF, Keshavarzian A, Shannon KM, Krajmalnik-Brown R, Wittung-Stafshede P, Knight R, Mazmanian SK. Gut Microbiota Regulate Motor Deficits and Neuroinflammation in a Model of Parkinson's Disease. Cell. 2016 Dec 1;167(6):1469-1480.e12. doi: 10.1016/j.cell.2016.11.018. PMID 27912057
- [Background] Frost F, Kacprowski T, Ruhlemann M, Pietzner M, Bang C, Franke A, Nauck M, Volker U, Volzke H, Dorr M, Baumbach J, Sendler M, Schulz C, Mayerle J, Weiss FU, Homuth G, Lerch MM. Long-term instability of the intestinal microbiome is associated with metabolic liver disease, low microbiota diversity, diabetes mellitus and impaired exocrine pancreatic function. Gut. 2021 Mar;70(3):522-530. doi: 10.1136/gutjnl-2020-322753. Epub 2020 Nov 9. PMID 33168600
- [Background] Yang J, Yang X, Wu G, Huang F, Shi X, Wei W, Zhang Y, Zhang H, Cheng L, Yu L, Shang J, Lv Y, Wang X, Zhai R, Li P, Cui B, Fang Y, Deng X, Tang S, Wang L, Yuan Q, Zhao L, Zhang F, Zhang C, Yuan H. Gut microbiota modulate distal symmetric polyneuropathy in patients with diabetes. Cell Metab. 2023 Sep 5;35(9):1548-1562.e7. doi: 10.1016/j.cmet.2023.06.010. Epub 2023 Jul 13. PMID 37451270
- [Background] Zhang T, Lu G, Zhao Z, Liu Y, Shen Q, Li P, Chen Y, Yin H, Wang H, Marcella C, Cui B, Cheng L, Ji G, Zhang F. Washed microbiota transplantation vs. manual fecal microbiota transplantation: clinical findings, animal studies and in vitro screening. Protein Cell. 2020 Apr;11(4):251-266. doi: 10.1007/s13238-019-00684-8. Epub 2020 Jan 9. PMID 31919742
- [Background] Lu G, Wang W, Li P, Wen Q, Cui B, Zhang F. Washed preparation of faecal microbiota changes the transplantation related safety, quantitative method and delivery. Microb Biotechnol. 2022 Sep;15(9):2439-2449. doi: 10.1111/1751-7915.14074. Epub 2022 May 16. PMID 35576458
- See also: The top 10 causes of death. World Health Organization. — http://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death
- See also: Diabetes Facts and Figures. International Diabetes Federation. — http://idf.org/about-diabetes/diabetes-facts-figures/